CLINICAL TRIAL: NCT04037124
Title: Oncological Outcome After Completing or Abandoning (Radical) Hysterectomy in Patients With Cervical Cancer and Intraoperative Detection of LN Positivity; ABRAX (ABandoning RAd Hyst in cerviX Cancer)
Brief Title: Oncological Outcome After Completing or Abandoning (Radical) Hysterectomy in Patients With Cervical Cancer and Intraoperative Detection of LN Positivity
Acronym: ABRAX
Status: Completed | Type: Observational
Sponsor: General University Hospital, Prague (Other)
Responsible Party: Principal Investigator, David Cibula, Head of Gynecologic Oncology Center, General University Hospital, Prague
Other Study IDs: ENGOT-Cx3/CEEGOG/ABRAX
Record Dates: First submitted 2019-07-21; First posted 2019-07-30 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Uterine Cervical Neoplasms
Keywords: Cervical cancer; Lymph node involvement; Radical hysterectomy; Radiotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cervical procedure abandoned: Cervical procedure (hysterectomy, radical hysterectomy or fertility sparing treatment) is abandoned due to intraoperatively reported lymph node matestasis. Patient is referred for primary (chemo)radiation.
- Cervical procedure completed: Cervical procedure (hysterectomy, radical hysterectomy or fertility sparing treatment) is completed. Patient is referred for adjuvant chemoradiation.
  Interventions: Procedure: Cervical procedure

INTERVENTIONS:
Procedure: Cervical procedure — simple hysterectomy, radical hysterectomy or fertility sparing surgery
  Groups: Cervical procedure completed

SUMMARY:
The ABRAX trial is multicentre retrospective cohort study. Included are patients with negative LN in clinical staging, in whom LN involvement is detected intraoperatively. Completion or abandonment of planned cervical procedure stratifies the cohort in two subgroups in which oncological outcome and morbidity will be compared.

The investigators hypothesise that in patients with intraoperative LN involvement, a completion of radical hysterectomy or other cervical procedure does not improve oncological outcome of definitive chemoradiation.

DETAILED DESCRIPTION:
The management of patients with intraoperative detection of lymph node (LN) involvement currently varies widely. Options include completing or abandoning radical hysterectomy, performing or abandoning pelvic lymph node dissection and even continuing with inframesenteric or infrarenal paraaortic lymph node dissection. The most significant aspect is the decision regarding the performance of radical hysterectomy, due to the high morbidity caused by combined treatment composed of radical parametrectomy and adjuvant radiotherapy in these patients - patients are referred to pelvic radiotherapy after distal ureters, bladder and rectum have been surgically dissected [1].

Data on the oncologic outcome of patients with LN involvement after radical hysterectomy and adjuvant radiotherapy are broadly available. Recent figures show five-year survival in stage IB at around 70-85 % [2,3]. In contrast, the data on patients in whom radical hysterectomy was abandoned due to intraoperative detection of LN involvement are scarce. Available literature mostly refers to small groups of cases with grossly involved LN detected during surgery [4-7].

The goal of this study is to obtain the best data available from an adequate number of patients treated by both types of management in the same period of time and to analyse the risks and benefits of the performance of radical hysterectomy if LN involvement is detected intraoperatively in spite of non-suspicious preoperative radiological assessment.

ABRAX is an international multicenter retrospective trial. Data of cervical cancer patients with preoperatively negative LN in whom nodal involvement is detected during operation will be evaluated. The protocol has been developed to be inclusive and reflect current clinical practice. All surgical approaches are eligible for the study. Lymph node infiltration can be detected either by intraoperative pathology assessment or by gross assessment (macroscopic suspicion has to be confirmed by the final histology). Sentinel or any other pelvic lymph node can be subject of intraoperative assessment. Any type of nodal metastasis (macrometastasis, micrometastasis ot isolated tumor cells) is considered a positive LN. All types of cervical procedures (such as conisation, simple hysterectomy, trachelectomy, any type radical hysterectomy or radical trachelectomy) are eligible for the trial and administration of neoadjuvant chemotherapy is not an exclusion criterion. The abandonment of planned cervical procedure depends solely on the decision of the surgeon and on local institutional guidelines. The completion or abandonment of cervical procedure stratifies the cohort in two subgroups.

The primary end-point is the progression free survival assessed separately in both subgroups. Prevalence of ≥ G2 treatment related morbidity (CTCAE), overall and pelvic progression free survival are the secondary end-points.

Oncological outcome will be stratified according to the prognostic parameters such as tumour size, number of involved LN, type of LN metastases, presence of LVSI (lymphovascular space invasion), tumor type, administration of neoadjuvant chemotherapy, performance of systematic pelvic lymphadenectomy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma, adenocarcinoma, adenosquamous carcinoma
* Stage pT1a - pT2b
* Patient referred for primary surgical treatment such as radical / simple hysterectomy or fertility-sparing procedure (FST) and LN staging
* Intraoperative detection of LN involvement (any type of metastasis):
* Macroscopic involvement = grossly involved lymph nodes (if confirmed by final pathology) OR Microscopic involvement = SLN / LN intraoperative pathologic evaluation (frozen section)
* Follow-up data available for ≥ 2 years
* Surgery performed between January 2005 and December 2015

Exclusion Criteria:

* Preoperative evidence of grossly involved LN
* Histologic subtypes other than those noted in the Inclusion criteria
* Negative pelvic LN
* LN involvement reported by the final histology but not detected during the surgery
* Unavailability of follow-up data

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Consecutive participant sampling of patients with pT1a - pT2b cervical cancer and no evidence of LN involvement in preoperative imaging who were referred for primary surgery with curative intent and in whom nodal involvement was discovered intraoperatively.
Sampling Method: Probability Sample
Enrollment: 718 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From date of surgery for cervical cancer until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 176 months
  Compare progression-free survival in cervical cancer patients in whom LN involvement was intraoperatively detected and in whom cervical procedure was completed vs. abandoned.

SECONDARY OUTCOMES:
Prevalence of treatment related morbidity | From date of surgery for cervical cancer until the date of last follow-up control or death from any cause, whichever came first, assessed up to 176 months
  Compare treatment related morbidity in cervical cancer patients in whom LN involvement was intraoperatively detected and in whom cervical procedure was completed vs. abandoned. Only adverse events ≥ grade 2 according to Common Terminology Criteria for Adverse Events (CTCAE) will be reported and evaluated.
Overall survival (OS) | From date of surgery for cervical cancer until the date of last follow-up control or death from any cause, whichever came first, assessed up to 176 months
  Compare overall survival in cervical cancer patients in whom LN involvement was intraoperatively detected and in whom cervical procedure was completed vs. abandoned.
Pelvic progression free survival | From date of surgery for cervical cancer until the date of first documented pelvic recurrence or date of death from any cause, whichever came first, assessed up to 176 months
  Compare pelvic progression-free survival in cervical cancer patients in whom LN involvement was intraoperatively detected and in whom cervical procedure was completed vs. abandoned.

CONTACTS AND LOCATIONS:
Locations (1):
- Gynecologic Oncology Center, Department of Obstetrics and Gynecology, First Faculty of Medicine, Charles University in Prague and General University Hospital in Prague, Czech Republic, Prague, MUDr., Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Landoni F, Maneo A, Colombo A, Placa F, Milani R, Perego P, Favini G, Ferri L, Mangioni C. Randomised study of radical surgery versus radiotherapy for stage Ib-IIa cervical cancer. Lancet. 1997 Aug 23;350(9077):535-40. doi: 10.1016/S0140-6736(97)02250-2. PMID 9284774
- [Background] Cibula D, Abu-Rustum NR, Dusek L, Zikan M, Zaal A, Sevcik L, Kenter GG, Querleu D, Jach R, Bats AS, Dyduch G, Graf P, Klat J, Lacheta J, Meijer CJ, Mery E, Verheijen R, Zweemer RP. Prognostic significance of low volume sentinel lymph node disease in early-stage cervical cancer. Gynecol Oncol. 2012 Mar;124(3):496-501. doi: 10.1016/j.ygyno.2011.11.037. Epub 2011 Nov 25. PMID 22120175
- [Background] Richard SD, Krivak TC, Castleberry A, Beriwal S, Kelley JL 3rd, Edwards RP, Sukumvanich P. Survival for stage IB cervical cancer with positive lymph node involvement: a comparison of completed vs. abandoned radical hysterectomy. Gynecol Oncol. 2008 Apr;109(1):43-8. doi: 10.1016/j.ygyno.2007.12.002. Epub 2008 Jan 29. PMID 18234297
- [Background] Potter ME, Alvarez RD, Shingleton HM, Soong SJ, Hatch KD. Early invasive cervical cancer with pelvic lymph node involvement: to complete or not to complete radical hysterectomy? Gynecol Oncol. 1990 Apr;37(1):78-81. doi: 10.1016/0090-8258(90)90312-9. PMID 2323617
- [Background] Bremer GL, van der Putten HW, Dunselman GA, de Haan J. Early stage cervical cancer: aborted versus completed radical hysterectomy. Eur J Obstet Gynecol Reprod Biol. 1992 Nov 19;47(2):147-51. doi: 10.1016/0028-2243(92)90045-z. PMID 1459328
- [Background] Suprasert P, Srisomboon J, Charoenkwan K, Siriaungul S, Khunamornpong S, Siriaree S, Phongnarisorn C, Lorvidhaya V. Outcomes of abandoned radical hysterectomy in patients with stages IB-IIA cervical cancer found to have positive nodes during the operation. Int J Gynecol Cancer. 2005 May-Jun;15(3):498-502. doi: 10.1111/j.1525-1438.2005.15315.x. PMID 15882176
- [Background] Gray HJ, Seifert E, Sal Y Rosas VG, Nicandri KF, Koh WJ, Goff BA. The abandoned radical hysterectomy for cervical cancer: clinical predictors and outcomes. Obstet Gynecol Int. 2010;2010:743794. doi: 10.1155/2010/743794. Epub 2010 Apr 28. PMID 20454444
- [Derived] Cibula D, Dostalek L, Hillemanns P, Scambia G, Jarkovsky J, Persson J, Raspagliesi F, Novak Z, Jaeger A, Capilna ME, Weinberger V, Klat J, Schmidt RL, Lopez A, Scibilia G, Pareja R, Kucukmetin A, Kreitner L, El-Balat A, Pereira GJR, Laufhutte S, Isla-Ortiz D, Toptas T, Gil-Ibanez B, Vergote I, Runnenbaum I. Completion of radical hysterectomy does not improve survival of patients with cervical cancer and intraoperatively detected lymph node involvement: ABRAX international retrospective cohort study. Eur J Cancer. 2021 Jan;143:88-100. doi: 10.1016/j.ejca.2020.10.037. Epub 2020 Dec 5. PMID 33290995
- [Derived] Dostalek L, Runnebaum I, Raspagliesi F, Vergote I, Dusek L, Jarkovsky J, Cibula D. Oncologic outcome after completing or abandoning (radical) hysterectomy in patients with cervical cancer and intraoperative detection of lymph node positivity; ABRAX (ABandoning RAd hyst in cerviX cancer). Int J Gynecol Cancer. 2020 Feb;30(2):261-264. doi: 10.1136/ijgc-2019-000890. Epub 2019 Nov 20. PMID 31748245